CLINICAL TRIAL: NCT04467684
Title: A Phase 1, Randomized, Double-Blind, Placebo Controlled, Dose-Escalation Study Investigating the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of CB-0406 Tablets in Healthy Volunteers
Brief Title: Study Investigating the Safety, Tolerability, and PK, PD, of CB-0406
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CB0406-12047
Record Dates: First submitted 2020-06-29; First posted 2020-07-13 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Healthy Volunteers
Keywords: single ascending dose (SAD); multiple ascending dose (MAD); CymaBay; CB-0406; arhalofenate; peroxisome proliferator-activated receptor gamma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The assignment to either CB-0406 or placebo will be blinded to the participants, investigators and staff at the study site. The pharmacy team will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort 1 (Experimental): Cohort 1: 100 mg CB-0406 (n=6)
  Interventions: Drug: CB-0406 100 mg
- Cohort 2 (Experimental): Cohort 2: 200 mg CB-0406 (n=6). Dose initiated following review of all safety data from Cohort 1 by a Safety Review Committee
  Interventions: Drug: CB-0406 200 mg
- Cohort 3 (Experimental): Cohort 3: 400 mg CB-0406 (n=6). Dose initiated following review of all safety data and PK data from Cohort 2 by a Safety Review Committee.
  Interventions: Drug: CB-0406 400 mg
- 800 mg (Experimental): Cohort 4: 800 mg CB-0406 (n=6). Dose initiated following review of all safety data and PK data from Cohort 3 by a Safety Review Committee.
  Interventions: Drug: CB-0406 800 mg
- 1000 mg (Experimental): Cohort 5: 1000 mg CB-0406 (n=6). Dose initiated following review of all safety data and PK data from Cohort 4 by a Safety Review Committee
  Interventions: Drug: CB-0406 1,000 mg
- Matched placebo (Placebo Comparator): Two subjects in each Cohort (1, 2, 3, 4, 5) are randomized to matched placebo
  Interventions: Drug: Matched placebo

INTERVENTIONS:
Drug: CB-0406 100 mg — Single oral dose
  Arms: Cohort 1
Drug: CB-0406 200 mg — Single oral dose
  Arms: Cohort 2
Drug: CB-0406 400 mg — Single oral dose
  Arms: Cohort 3
Drug: CB-0406 800 mg — Single oral dose
  Arms: 800 mg
Drug: CB-0406 1,000 mg — Single oral dose
  Arms: 1000 mg
Drug: Matched placebo — Color and size matched placebo
  Arms: Matched placebo

SUMMARY:
The study is designed as a single center, randomized, double-blind, placebo-controlled study to assess the PK, safety, tolerability and PD of CB-0406 in healthy participants. The study will be conducted as a 2-part study.

DETAILED DESCRIPTION:
The study is designed as a 2-part study:

Part 1 is designed as single ascending dose (SAD) escalation study investigating 5 dose levels. Each cohort will consist of participants (N=8) to be randomly assigned to receive a blinded oral dose of CB-0406 (n=6) or placebo (n=2). Dose levels of CB-0406 in the sequential cohorts will be 100 mg, 200 mg, 400 mg, 800 mg or 1000 mg to be administered once on each cohorts study Day 1.

Part 2 is designed as multiple ascending dose (MAD) escalation study investigating up to 5 dose levels as determined by the SAD cohort. Doses will be determined following completion and review of the safety and PK findings for Cohorts 1 to Cohort 5 in Part 1.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for study entry participants must satisfy all of the following criteria:

1. Provide written informed consent before any study specific evaluation is performed;
2. Healthy adult male and female volunteers between the ages of 18 and 65 years, inclusive, at screening;
3. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

   * Not of childbearing potential, defined as surgically sterile (documented hysterectomy, bilateral salpingectomy, tubal ligation or bilateral oophorectomy - verbal confirmation through medical history review acceptable) or postmenopausal (no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy; however, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient);
   * Of childbearing potential and agrees to use a highly effective method of contraception consistently during the treatment period and for at least 30 days after the dose of study treatment;
4. A male patient with a female partner of childbearing potential is eligible to participate if he and his female partner agrees to use acceptable contraception during the treatment period and for at least 30 days after the last dose of study treatment and refrains from donating sperm during this period.
5. Body mass index of 18.0 to 32.0 kg/m2, inclusive, at screening;
6. Hematology, clinical chemistry, coagulation and urinalysis test results within normal ranges or has no clinically relevant deviations, as determined by the investigator in consultation with sponsor, at screening and Day -1. Tests with out of range values at screening or Day -1 may be repeated once per assessment point;
7. No clinically significant abnormalities noted in medical history; or discovered by physical examination, ECG assessment, or measurement of vital signs at screening and Day -1;
8. Able and willing to abstain from alcohol, caffeine or caffeine-containing products, grapefruit or grapefruit juice, St John's wort, and herbal supplements for from 24 hours before Day -1 until the end of the confinement period and for 24 hours prior to additional visits to the study site.
9. Agree to not engage in heavy exercise (e.g., marathon runners, weight-lifting) within 1 week prior to dosing until the final study visit.
10. Able and willing to comply with the protocol and study procedures;

Exclusion Criteria:

Participants will be excluded from the study if one or more of the following criterion are applicable:

1. Has an active or recurring clinically significant disorder of the skin, head, ears, eyes, nose, or throat; an active or recurring clinically significant disorder of the respiratory, cardiovascular, gastrointestinal, endocrine/metabolic, genitourinary, neurologic, hematologic, musculoskeletal, immunologic, or psychological/psychiatric system; or a disease requiring medical treatment;
2. Previous history of any surgical or medical condition that might significantly alter the absorption, distribution, metabolism, or excretion of CB-0406, such as stomach or intestinal surgery or resection (e.g., gastrectomy or any type of gastric by-pass surgery or gastric banding procedure);
3. Planning any elective medical treatment or surgery during the trial period or within 30 days of Day -1;
4. Any evidence or treatment of malignancy (other than localized basal cell cancer, squamous cell skin cancer, or cancer in situ that has been resected) within the previous 5 years;
5. Known history of allergic reactions to or have previously received arhalofenate, MBX-102, JNJ39659100, Metaglidasen, and/or K 118;
6. Previous history or evidence at screening of sick sinus syndrome or second- or third-degree atrioventricular block or any cardiac arrhythmia other than a benign sinus arrhythmia. Participant has not had a myocardial infarction within the last 6 months;
7. Clinically significant renal disease, nephrectomy, renal transplant or estimated glomerular filtration rate of <90 mL/min/1.73 m2 at screening based on Chronic Kidney Disease Epidemiology Collaboration creatinine equation (2009).
8. Blood pressure after resting for at least 5 minutes that is higher than 150 mm Hg systolic or 95 mm Hg diastolic, or lower than 90 mm Hg systolic or 50 mm Hg diastolic at screening or Day -1. A single repeat measurement at screening or Day -1 is allowed based on the investigator's judgment;
9. Pulse rate obtained from vital signs after resting for 5 minutes that is outside the range of 45 to 90 beats per minute at screening or Day -1. A single repeat measurement is allowed at screening and Day -1 for eligibility based on the investigator's judgment;
10. History of drug or alcohol abuse within the last 2 years;
11. Positive screen for drugs of abuse (amphetamines, methamphetamines, methadone, barbiturates, benzodiazepines, cocaine, opiates, methylenedioxymethamphetamine, phencyclidine, tetrahydrocannabinol), tricyclic antidepressants, cotinine or alcohol at screening or Day -1;
12. Smoke more than 2 cigarettes per week and have a positive cotinine test at screening or Day -1. Participants must agree to refrain from smoking from 24 hours prior to Day -1 until completion of the end of study (EOS) visit.
13. Used or are using prescription or over-the-counter medications, dietary/nutritional supplements (except for multivitamins at the recommended dose and paracetamol, up to 2g in any one day) within 14 days prior to Day 1 and for the duration of the trial.
14. Received an investigational drug within 30 days or 5 half -lives (whichever is longer) prior to Day 1.
15. Donated more than 450 mL of blood within 30 days prior to Day 1;
16. Evidence of clinically significant hepatic impairment including alanine aminotransferase or aspartate aminotransferase >1.5 times the upper limit of normal, with the exception of elevated bilirubin due to Gilbert's syndrome based on bilirubin fractionation at screening;
17. Positive test result at screening for human immunodeficiency virus (Types 1 or 2) antibody, hepatitis B surface antigen, or hepatitis C virus antibody;
18. Clinically significant acute illness within 4 weeks or other illness deemed to be significant by investigator with agreement of sponsor within 5 days before Day 1;
19. Participant or a family member of the participant is a member of the professional or ancillary personnel working at the investigative site involved in the study;
20. Participant, in the opinion of the investigator, should not participate in the study;
21. Participant has received blood products within 2 months prior to Day -1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Parameters | Part 1: Day 1 to Day 15; Part 2: Day 14 to Day 28
  Concentration of CB-0406 in plasma.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Part 1: Day 1 to Day 22; Part 2: Day 1 to Day 35
  Incidence of adverse events
Pharmacodynamic Activity | Part 1: Day 1 to Day 15; Part 2: Day 14 to Day 28
  Evaluation of relative changes from baseline in plasma IL-1β and serum urate over time
Incidence of abnormal laboratory tests results | Part 1: Screening, Day -1, Day 2, Day 4, Day 9, Day 15, EOS/ET Part 2: Screening, Day -1, Day 2 to 13, Day 14, Day 16, Day 20, Day 28, EOS/ET
  Evaluation of clinically significant changes from baseline in laboratory evaluation (hematology, chemistry, coagulation, urinalysis)
Incidence of Abnormal Vital Signs | Part 1: Every visit; Part 2 Every visit
  Evaluation of clinically significant changes in vital signs will include body temperature (tympanic), respiratory rate, heart rate and systolic and diastolic blood pressure
Incidence of Abnormal ECGs | Part 1: Screening, Day 1, Day 2, Day 3, Day 4, Day 9, Day 15, EOS/ET; Part 2 Screening, Day 1, Day 2 to 13, Day 14, Day 16, Day 20, Day 28, Day 35
  The following parameters will be assessed using a 12-lead ECG: heart rate, PR, QRS, QT, QTcF (Fridericia's formula).
Incidence of Abnormal Physical Exams | Part 1: Day -1 and at the EOS/ET visit; Part 2 Screening, Day 1, Day 2 to 13, Day 4, Day 16, Day 20, Day 28, EOS/ET
  Assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Watkins, DO, MSPH, Study Director — Gilead Sciences
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aronow WS, Harding PR, Khursheed M, Vangrow JS, Papageorge's NP, Mays J. Effect of halofenate on serum lipids. Clin Pharmacol Ther. 1973 May-Jun;14(3):358-65. doi: 10.1002/cpt1973143358. No abstract available. PMID 4572798
- [Background] Dujovne CA, Azarnoff DL, Pentikainen P, Manion C, Hurwitz A, Hassanein K. A two-year crossover therapeutic trial with halofenate and clofibrate. Am J Med Sci. 1976 Nov-Dec;272(3):277-84. doi: 10.1097/00000441-197611000-00005. PMID 797258
- See also: CymaBay Therapeutics — http://www.cymabay.com/